CLINICAL TRIAL: NCT07214493
Title: Impact of a Prosthetic Foot With Adjustable Heel Height on Physical Appearance and Participation: a Randomized Crossover Trial.
Brief Title: Study on a Prosthetic Foot With Adjustable Heel Height
Acronym: ADJUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock France SNC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BP-11-PT009
Record Dates: First submitted 2025-09-23; First posted 2025-10-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lower Limb Amputation Above Knee; Lower Limb Amputation Below Knee
Keywords: Lower limb amputation; Prosthetic foot; Adjustable heel height; Hydraulic ankle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taleo Adjust foot then usual foot (Other): The participant is first fitted with the Taleo Adjust foot for 30 days, then is fitted with their usual foot for 30 days.
  Interventions: Device: Taleo Adjust; Device: The usual participant's foot
- Usual foot then taleo Adjust foot (Other): The participant is first fitted with their usual foot for 30 days, then fitted with the Taleo Adjust foot for 30 days
  Interventions: Device: Taleo Adjust; Device: The usual participant's foot

INTERVENTIONS:
Device: Taleo Adjust — The Taleo Adjust foot is an energy-storage-and-return (ESR) prosthetic foot with a hydraulic ankle joint that allows an adjustable heel height from 0 to 7 cm.
Device: The usual participant's foot — The usual foot of the participant is an Energy Storage and Return (ESR) prosthetic foot (no heel height adjustement)

SUMMARY:
Most prosthetic feet have a fixed heel height, which requires users to always wear shoes with the same heel height. A fixed heel height is a significant constraint, whereas the ability to choose one's clothing freely is an important aspect of coping with a physical disability.

The Taleo Adjust is a prosthetic foot with a hydraulic ankle that allows the user to adjust the heel height from 0 to 7 cm, depending on the type of shoe worn.

This study aims to evaluate the impact of an adjustable-heel-height foot on physical appearance and participation.

DETAILED DESCRIPTION:
The amputation or absence of a lower limb affects both mobility and appearance, which can lead to restrictions in social, family, and professional participation. The choice of prosthetic components aims to compensate as effectively as possible for the functional and physical disability, in line with the patient's expectations and life plan.

The prosthetic foot is a key component of the prosthesis. Most feet have a fixed heel height-most often around 10 to 15 mm-which requires users to always wear shoes with the same heel height, since prosthetic alignment, essential for harmonious and safe walking, is set accordingly.

A fixed heel height is a significant constraint for many users who wish to wear different types of shoes for aesthetic reasons (e.g., city shoes or pumps for work or going out; flip-flops or flat ballet flats in summer), for safety reasons (e.g., boots for motorcycling or gardening), or to be able to walk barefoot (e.g., at home). The ability to choose one's clothing freely is an important aspect of coping with a physical disability.

The Taleo Adjust is an energy-storing and energy-returning prosthetic foot with a hydraulic ankle that allows the user to adjust the heel height from 0 to 7 cm, depending on the type of shoe worn. Thanks to this articulation, prosthetic alignment is preserved and walking quality is not compromised.

This study aims to evaluate the impact of an adjustable-heel-height foot on physical appearance and participation.

ELIGIBILITY:
Inclusion Criteria :

* Adult patient with a major lower limb amputation whose life project includes:
* movement in buildings other than the home (ICF d4601),
* movement outside the home and other buildings (ICF d4602),
* and other specified activities related to movement in other various places (ICF d4608).
* Patient who has been using an Enregy storage and Return (ESR) foot for at least 3 months
* Patient who wishes to walk with shoes with different heel heights, and/or barefoot

Exclusion Criteria:

* Patient with a high impact level (e.g.: sport)
* Patient with hip disarticulation or equivalent
* Patient with an unstabilised residual limb and/or an unsuitable socket
* Patient who cannot be fitted with a Taleo Adjust foot due to the technical characteristics of the product (user weight greater than 115kg; required foot size <22 or >28; mounting height less than 118 mm)
* Patient whose usual foot has a heel height adjustment system
* Patient unavailable for the duration of the study and/or unable to understand the instructions and/or answer questionnaires in French
* Patient already participating in another study
* Patient in an emergency situation or pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Evaluation Questionnaire - Appearance scale (PEQ-AP) | 30 days
  A 5-item self-reported measure of the appearance domain. The participant rates each item by marking a 100-mm line. Scores range from 0 to 100, with higher scores indicating a more positive perception.

SECONDARY OUTCOMES:
Patient Specific functional Scale (PSFS) | 30 days
  A self-reported measure of participation based on 3 to 5 self-selected activities that the participant cannot perform or can perform only with difficulty. Participants will be asked to rate their ability to perform each activity on a numerical scale from 0 (unable to perform the activity) to 10 (able to fully perform the activity).
Psychosocial Impact of Assistive Device Scale (PIADS) | 30 days
  A 26-item questionnaire that assesses the effects of an assistive device on functional independence, well-being, and quality of life from the perspective of the person's disability. Each item is rated on a 7-point Likert scale ranging from -3 (maximum negative impact) to +3 (maximum positive impact).
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | 30 days
  A 12-item self-reported measure of the participant's satisfaction with the device's technology and the services associated with it. An average satisfaction rating can be calculated on a scale from 1 to 5, with 1 = "Not at all satisfied" and 5 = "Very satisfied". A higher score indicates greater satisfaction. It also allows the participant to express the three criteria that are most important to them.
Visual Analog Scale (VAS) for the adequacy to life's project | 30 days
  An 11-level numerical scale ranging from 0 (total dissatisfaction) to 10 (total satisfaction), measuring how well the device aligns with the participant's life project
EuroQuol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 30 days
  A self-reported measure of health status composed of five dimensions: mobility, self-care, ability to perform usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-point scale. A utility index, which is a single value derived from a patient's responses to these dimensions, can be calculated using a population-specific value set, typically ranging from 0 (death) to 1 (perfect health).
  Health status is also expressed using the EQ-VAS (Visual Analog Scale). The EQ-VAS records the patient's self-assessment of health on a vertical visual analog scale, ranging from 0 "The worst health you could imagine" to 100 "The best health you could imagine."
Prosthetic Limb Users Survey of Mobility (PLUS-M) | 30 days
  A 12-items self-reported measure of mobility as the ability to move intentionally and independantly from one place to another. Questions cover movements that range from basic ambulation to complex activities . Response options going from 1 (unable to do) to 5 (without any difficulty), reflecting the degree of difficulty with which respondents report they can perform these activities. The PLUS-M™ 12-item short form provides a T-score ranging from 21.8 to 71.4, with higher scores indicating better mobility.
Socket Comfort Scale (SCS) | 30 days
  A 11-levels numerical scale going from 0 (the most uncomfortable socket) to 10 (the most comfortable socket), measuring the perceived comfort in the socket.

CONTACTS AND LOCATIONS:
Overall Officials: Brice LAVRARD, Dr., Study Chair — Institut Merle d'Aubigné - VALENTON; Isabelle LOIRET, Study Chair — IRR Louis Pierquin - NANCY
Locations (5):
- France (5):
  - CH Cornouaille, Concarneau
  - CHU Grenoble, Échirolles
  - IRR Louis Pierquin, Nancy
  - CRRF La Tourmaline, Saint-Herblain
  - Institut Merle d'Aubigné, Valenton

IPD SHARING:
Plan to Share IPD: No